CLINICAL TRIAL: NCT04662827
Title: The Effect of Palmitylethanolamide on Central and Peripheral Sensitization After Heat-induced Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1403/2019
Record Dates: First submitted 2020-11-23; First posted 2020-12-10 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Pain, Chronic; Pain, Acute; Central Sensitisation; Neuroinflammatory Response
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: doubleblind, placebo-controlled,prospective crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking is done by the pharmacological department also produces the placebos
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palmithylethanolamid (Experimental): Probands receive PEA 3xday for 28 days, 8 weeks wash out will follow, then they receive placebo for 28 days
  Interventions: Dietary Supplement: Palmithylethanolamid; Other: placebo
- placebo (Placebo Comparator): Probands receive placebo 3xday for 28 days, 8 weeks washout will follow, then they receive PEA for 28 days
  Interventions: Dietary Supplement: Palmithylethanolamid; Other: placebo

INTERVENTIONS:
Dietary Supplement: Palmithylethanolamid — PEA 3x/d
Other: placebo — placebo 3x/d

SUMMARY:
This planned study is based on a randomized, placebo-controlled cross-over design.

Palmityhlethanolamide (PEA) is an endogenous fatty acid amide from the group of N-Acetylethanolamides, which analgesic, anti-inflammatory and neuroprotective effects can be attributed to this. In clinical studies, PEA has mainly been used as an adjuvant in pain therapy. The previous data show clinical efficacy without conclusions that can be drawn about the underlying mechanisms - these have not yet been investigated in a human experiment.

The planned study, which demonstrates the mode of action of PEA using an established pain model on healthy volunteers, will help to assign the efficacy to peripheral or central nervous systems. These mechanisms allow to establish mechanism-oriented therapy approaches. These findings are essential for a better understanding of the clinical efficacy and to evaluate the correct fields of application.

DETAILED DESCRIPTION:
Palmityhlethanolamide (PEA) is an endogenous fatty acid amide from the group of N-Acetylethanolamides, which analgesic, anti-inflammatory and neuroprotective effects can be attributed to this. It is referred to as "dietary Food for special medical purposes". Different mechanisms of action have been described, including an effect on mast cells, ATP-sensitive K channels and TRP channels. In an animal study in mice it could be shown that the antinociceptive properties of PEA can be blocked by a CB2-cannabinoid antagonist. Overall, PEA seems to play a relevant role in the body's own regulation of neurogenic inflammation.

In clinical studies, PEA has mainly been used as an adjuvant in pain therapy. In a recent metaanalysis of studies in which PEA was used to treatment of neuropathic or chronic pain, a significant effect can be shown. Remarkably none of the 1188 patients who took PEA for up to 60 days had reported side effects.

"Repetitive phasic heat application" is a validated method to generate a short-term peripheral and central sensitization. As a non-invasive human pain model, it is therefore well suited to examine analgesic and antihyperalgesic effects of pharmaceuticals.

The data of the above meta-analysis show clinical efficacy without conclusions that can be drawn about the underlying mechanisms - these have not yet been investigated in a human experiment. Our planned study, which demonstrates the mode of action of PEA using an established pain model on healthy volunteers, will help to assign the efficacy to peripheral or central nervous systems. These mechanisms allow to establish mechanism-oriented therapy approaches. These findings are essential for a better understanding of the clinical efficacy and to evaluate the correct fields of applikation. If there is peripheral efficacy, this would qualify PEA for use in acute pain. However, if the effect is explained by central mechanisms, PEA can be useful in the area of chronic pain, and also in neuropathic pain. Accordingly, the results of this experimental human study are groundbreaking for the planning of future application studies or clinical use.

Questions:

In this study four questions were to be answered:

1. Can spontaneous pain after repetitive phasic heat application be reduced by the intake of PEA?
2. Can central sensitization be influenced by the intake of PEA?
3. Can peripheral sensitization be influenced by the intake of PEA?
4. Can the endogenous pain inhibition be influenced by the intake of PEA?

The following methods are used to answer these questions.

1. Spontaneous pain is measured using Visual Analog Scale (VAS).
2. To assign an effect to central sensitization, the sensitivity to mechanical stimuli, i.e. Pinprick hyperalgesia or allodynia is the established marker.
3. Efficacy on peripheral sensitization can be assessed by measuring the heat- thresholds.
4. The endogenous pain inhibition is tested by the examination of the "conditioned pain modulation".

Hypotheses

Null hypothesis:

Taking PEA 3x400mg for 28 days changes, compared to placebo spontaneous pain after repetitive phasic heat application.

Alternative hypothesis:

Taking PEA 3x400mg for 28 days changes, compared to placebo spontaneous pain after repetitive phasic heat application.

Secondary hypotheses:

There is a significant difference in the size of mechanical allodynia distance after repetitive phasic heat application compared to placebo intake.

PEA induces a change in Pinprick hyperalgesia compared to placebo after repetitive phasic heat application.

PEA induces a change in thermal perception and pain threshold compared to placebo after repetitive phasic heat application.

PEA induces a change in "conditioned pain modulation" compared to placebo.

Method:

This study is based on a randomized, placebo-controlled cross-over design. The patients take either the test substance or placebo for 28 days according to a randomization generated via "randomizer.at". Both the patients and the study staff responsible for collecting the measurement parameters are blinded by the order in which the tablets are taken, as the individual tablets are stored in doses that are only marked with a code, that does not allow to identify whether they are verum or placebo preparations. A staff member not participating in the study will dissolve the code at the end of the study.

After recruitment, information and inclusion of the subjects in the study, the first baseline measurement is performed. This is followed by randomization into 2 groups. After 28 days, during which either the verum or study substance is taken, the influence on the "conditioned pain modulation" is measured. The repetitive phasic heat application according to the published procedures follows. A 3x3cm area on the volar forearm is heated repeatedly using a TSA-II NeuroSensoryAnalyser. The thermode starts at 32.0°C and heats up to 48.0°C at 10°C/sec and cools down to 32.0°C after 6 seconds. This is repeated 6 times in total. This is followed by a 30 second pause and then 6 more heatings. A total of 10 blocks with 6 heatings each are performed.

At the end of the last block, spontaneous pain is determined using the Visual Analogue Scale.

Since primary and secondary hyperalgesia is most pronounced at 1 hour after repetitive phasic heat application, 60 minutes after the last heating, the measurement of allodynia distance and pinprick hyperalgesia is performed in immediate temporal sequence and the heat pain and perception threshold is determined.

After an 8-week wash-out phase, a new baseline measurement is taken before the other substance is taken for 28 days. This is followed by a new examination of the conditioned pain modulation, a repetitive phasic heat application and the recording of the measurement parameters according to the sequence described above.

Statistics:

In cooperation with the Institute for Medical Informatics, Statistics and Documentation of the Medical University of Graz, the T-test for paired samples was defined for biometric planning, the planned evaluation is based on a linear mixed model.

Study substance The volunteers will each receive 90 tablets containing either palmitoylethanolamide 400mg (OptiPEA.) or an optically identical placebo manufactured by our institutional pharmacy. The study substance is supplied by the company Innexus Nutraceuticals. It is taken at 8-hour intervals. The last dose is taken in the morning before the study visit. To increase the adherence to the therapy, an electronic reminder is given via cell phone.

Parameter

Spontaneous pain:

Directly after the last heat application, the spontaneous pain is recorded using the VAS scale, which is used throughout the LKH Univ.-Klinikum Graz.

Allodynia:

Starting from the center of the thermal application, a von Frey filament (128 mN) is applied to the skin in 4 radial lines at a 5 mm interval, first from the inside to the outside, then from the outside to the inside, and the distance at which an unpleasant pointed sensation first occurs is determined. The 8 measurements are averaged.

Pinprick hyperalgesia:

By means of a pinprick with 256 mN a pointed stimulus is applied. The test site is 5 cm proximal to the center of the thermal stimulation area. A numerical scale (0-100) is used to measure how painful this stimulus is.

Heat pain and perception threshold:

The heat detection threshold and the heat pain threshold are determined according to the guidelines of the German Research Association for Neuropathic Pain, which involves heating the skin with TSA-II NeuroSensoryAnalyser. The test person can stop the heatig by pressing a stop button. This should be done at the first time he/she notices that the skin is warming up (heat detection threshold) or at the time he/she notices a pulling, burning or pricking sensation in addition to the feeling of heat (heat pain threshold). The measurements are taken 3 times each and the results are averaged.

Conditioned pain modulation Conditioned pain modulation describes the function of the descending, pain-inhibiting system. First, the force with which pressure on the adductor pollicis brevis muscle of the non-dominant hand is not only perceived as pressure, but also as a stabbing, burning or pulling sensation is determined using a pressure gauge. Subsequently, the contralateral hand is immersed in ice water until the subject feels a pain intensity of NRS 40 (101-part scale). The pressure pain threshold is then immediately raised again.

Adverse effects:

Possible adverse effects are assessed and documented at each study visit. In addition, the subjects are informed about the necessity of immediate telephone contact in case of the occurrence of undesirable side effects.

Sample Size The sample size was calculated by Mag. Schwantzer, Institute for Medical Informatics, Statistics and Documentation (IMI), Medical University of Graz. The database was based on the study by Jurgens et al, in which repetitive phasic heat application was tested in healthy volunteers.

In this publication, the mean value for maximum pain was 72.2, the standard deviation was given as 5.4. Assuming more conservative baseline numbers for case number estimation (SD=10.8), a sample size of 12 on a paired sample T-test with alpha=5% would have 80% power to detect a difference of 10 VAS units. To compensate for any drop-outs, a sample size of 14 subjects is included in the study. Statistical evaluation is performed by the T-test for paired samples or the Wilcoxon sign test, depending on the central tendency.

Recruitment of test persons / education Recruitment is done by posting on notice boards at the ÖH an der KF-Uni Graz (main building, Resowi, Wall building).

Subjects are asked orally whether they participate in another study at the same time or whether a required period of time has elapsed since participation in another study. They confirm this with their signature.

An anesthesiologist involved in the study will provide the information. Consent is then given by signing a written information sheet.

PEA is sold as "dietary food for special medical purposes". In a recent literature analysis, no side effects were reported in 1188 patients who took PEA for up to 60 days. Nevertheless, the company Innexus Nutraceuticals describes in an information leaflet that PEA "slows down intestinal function". Some people may suffer from constipation or a feeling of fullness as a result".

The investigation of pain and perception thresholds according to the specifications of the "German Research Association for Neuropathic Pain" is an established procedure in both human research and clinical investigation. No danger is to be expected for the individual test person.

The application of "repetitive phasic heat application" is an established human pain model. The maximum heat exposure of 48°C does not lead to skin damage. The changes in pain sensitivity are locally very limited and normalize within a few hours.

If the individual test person is willing to be exposed to a pain stimulus for a limited period of time, there is no foreseeable risk for him/her.

ELIGIBILITY:
Exclusion Criteria:

* Chronic pain
* Analgesic intake
* Neurological illness
* Dermatological illness
* Cardiovascular illness
* PEA Allergy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Change in spontaneous pain intensity | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 112 before repeated heat application -->Day 112 1 hour after repeated heat application
  is measured on a visual analogue scale (0 means no pain and 10 means the worst imaginable pain)
Change in Allodynia | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 112 before repeated heat application -->Day 112 1 hour after repeated heat application
  measured in radial distance in mm
Change in Hyperalgesia | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 112 before repeated heat application -->Day 112 1 hour after repeated heat application
  measured with pinpricks, that are preset different peak stimulus. A numerical scale (0-100) is used to measure how painful the stimulus is.
Change in heat detection threshold | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 112 before repeated heat application -->Day 112 1 hour after repeated heat application
  measured in degrees
Change in heat pain threshold | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 112 before repeated heat application -->Day 112 1 hour after repeated heat application
  measured in degrees
Change in conditioned pain modulation | -->Day 0 -->Day 28 before repeated heat application -->Day 28 1 hour after repeated heat application --> Day 56 -->Day 112 before repeated heat application -->Day 112 1 hour after repeated heat application
  measures the descending analgesic System with the help of a pressure agometer in kg

CONTACTS AND LOCATIONS:
Overall Officials: helmar Boremann-cimenti, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Medical University of Graz, Graz, Austria. helmar.bornemann@medunigraz.at
Locations (1):
- Medical university of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paladini A, Fusco M, Cenacchi T, Schievano C, Piroli A, Varrassi G. Palmitoylethanolamide, a Special Food for Medical Purposes, in the Treatment of Chronic Pain: A Pooled Data Meta-analysis. Pain Physician. 2016 Feb;19(2):11-24. PMID 26815246